CLINICAL TRIAL: NCT01179360
Title: Clinical Value of Combined [18F]Fluoro-2-deoxy-D-glucose (FDG) PET/CT Imaging in Response Evaluation After Radiochemotherapy in Patients With Potentially Operable Locally Advanced Head and Neck Squamous Cell Carcinoma.
Brief Title: Combined FDG PET/CT Imaging in Response Evaluation After Radiochemotherapy in Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Acronym: ECLYPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Tim Van den Wyngaert, Senior consultant, University Hospital, Antwerp
Other Study IDs: IWT-90867
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Locally Advanced Squamous Cell Carcinoma of the Head and Neck Region
Keywords: Locally advanced; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Imaging group
  Interventions: Other: Integrated FDG PET/CT

INTERVENTIONS:
Other: Integrated FDG PET/CT — Optimized PET/CT imaging with dedicated head-and-neck protocol

SUMMARY:
To determine if combined [18F]fluoro-2-deoxy-D-glucose (FDG) positron emission tomography/computed tomography (PET/CT) is performant enough with respect to detecting residual lymph node involvement after chemoradiation in order to omit planned neck dissections in patients with locally advanced potentially operable, N2 and N3 head and neck squamous cell carcinoma (HNSCC).

Primary study hypothesis: The lower bound of the 95% confidence interval (CI) of the negative predictive value (NPV) of FDG PET/CT to detect residual malignant lymph node involvement at 12 weeks after completing chemoradiation will exceed 85%.

DETAILED DESCRIPTION:
Patients with locally advanced, N2 and N3 head and neck squamous cell carcinoma (HNSCC) will be recruited. All subjects receiving induction chemotherapy will undergo a baseline integrated [18F]fluoro-2-deoxy-D-glucose (FDG) positron emission tomography/computed tomography (PET/CT) scan before the start of concurrent chemoradiation. This baseline assessment is optional in patients not receiving neo-adjuvant treatment.

All patients will undergo a dedicated FDG PET/CT protocol 12 weeks after the end of chemoradiation (primary endpoint). In PET/CT negative patients, 2 monthly control visits will be performed complemented with additional imaging as required. All patients will undergo PET/CT 1 year after completing chemoradiation unless recurrent/residual disease was already proven pathologically. Patients with a PET/CT suspected for residual nodal disease must have pathological proof of nodal involvement (fine needle aspiration in non-operable patients or neck dissection in the others) before salvage chemotherapy is started.

In a subset of patients receiving induction chemotherapy prior to concurrent chemoradiation, an additional FDG PET/CT scan will be performed at baseline and after 1 cycle of chemotherapy to evaluate the metabolic response to the treatment (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Patients with locoregionally advanced HNSCC (clinically and/or radiological N2 or N3 disease, any T stage) with no evidence of distant metastases, scheduled for concurrent chemoradiation and being potential candidates for a subsequent neck dissection.
* Induction chemotherapy is allowed if this approach is followed by concurrent chemo-radiation.

Exclusion Criteria:

* Other head and neck cancer histologies
* Upfront inoperable patients in the neck (eg. carotid invasion)
* Presence of distant metastases
* A history of another primary malignancy, except when disease-free for at least 5 years after radical treatment, or except for treated basaloid skin cancer or in situ carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced, N2 and N3 HNSCC
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2011-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Negative predictive value (NPV) of FDG PET/CT | 12 weeks after chemoradiation
  The negative predictive value (NPV) of FDG PET/CT for detecting residual nodal involvement

SECONDARY OUTCOMES:
The sensitivity and specificity of high-resolution FDG PET/CT | 12 weeks after chemoradiation
The sensitivity and specificity of dual time point FDG PET/CT | 12 weeks after chemoradiation
The number of additional metastases found on PET and the % change in patient management | Prior to start of chemoradiation
DFS and OS, correlation with baseline SUV, early PET response and with HPV status | 1 year after completion of chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Stroobants, MD, PhD, Principal Investigator — University Hospital, Antwerp; Laurens Carp, MD, Principal Investigator — University Hospital, Antwerp
Locations (3):
- Belgium (2):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Turnhout, Turnhout, Antwerp
- Academisch Ziekenhuis Vrije Universiteit Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Result] Van den Wyngaert T, Helsen N, Carp L, Hakim S, Martens MJ, Hutsebaut I, Debruyne PR, Maes ALM, van Dinther J, Van Laer CG, Hoekstra OS, De Bree R, Meersschout SAE, Lenssen O, Vermorken JB, Van den Weyngaert D, Stroobants S; ECLYPS investigators. Fluorodeoxyglucose-Positron Emission Tomography/Computed Tomography After Concurrent Chemoradiotherapy in Locally Advanced Head-and-Neck Squamous Cell Cancer: The ECLYPS Study. J Clin Oncol. 2017 Oct 20;35(30):3458-3464. doi: 10.1200/JCO.2017.73.5845. Epub 2017 Aug 30. PMID 28854069
- [Derived] Helsen N, Van den Wyngaert T, Carp L, De Bree R, VanderVeken OM, De Geeter F, Maes A, Cambier JP, Spaepen K, Martens M, Hakim S, Beels L, Hoekstra OS, Van den Weyngaert D, Stroobants S; ECLYPS Consortium; Van Laer C, Specenier P, Maes A, Debruyne P, Hutsebaut I, Van Dinter J, Homans F, Goethals L, Lenssen O, Deben K. Quantification of 18F-fluorodeoxyglucose uptake to detect residual nodal disease in locally advanced head and neck squamous cell carcinoma after chemoradiotherapy: results from the ECLYPS study. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1075-1082. doi: 10.1007/s00259-020-04710-4. Epub 2020 Feb 10. PMID 32040611